CLINICAL TRIAL: NCT00092001
Title: A Phase 2 Efficacy And Safety Study Of SU011248 In Patients With Metastatic Non-Small Cell Lung Cancer
Brief Title: Study Of SU011248 In Patients With Metastatic Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer Inc
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A6181040
Record Dates: First submitted 2004-09-21; First posted 2004-09-27 (Estimated); Last update posted 2008-10-16 (Estimated); Status verified 2008-10

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Non-small cell lung cancer, carcinoma, sunitinib, Phase 2
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Carcinoma | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Sunitinib

INTERVENTIONS:
Drug: Sunitinib — Sunitinib 50 mg by oral capsule daily for 4 weeks in every 6 week cycle until progression or unacceptable toxicity.
  Other Names: Sutent, SU011248

SUMMARY:
The purpose of this study is to test whether SU011248 has activity and is safe in patients with metastatic non-small cell lung cancer (NSCLC) who have failed a platinum-containing regimen and docetaxel.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed advanced or metastatic Non-Small Cell Lung Cancer that cannot be cured with surgery, radiation, or combination thereof
* No more than 2 prior chemotherapy treatments including treatment with a platinum containing therapy
* Evidence of measurable disease by radiographic technique
* Male or Female, 18 years or older
* ECOG performance status of 0 or 1
* Resolution of all acute toxicities of prior therapies
* Adequate organ function

Exclusion Criteria:

* Major surgery or radiation therapy within 4 weeks
* Severe hemorrhage within 4 weeks
* Previous treatment with anti-angiogenesis agents
* Diagnosis of second malignancy within last five 5 years
* History of or known brain metastases, spinal cord compression, or carcinomatous meningitis
* Known HIV
* Serious acute or chronic illness
* Current treatment on another clinical trial
* Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2005-01; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Overall confirmed objective response rate (ORR) | From screening until at least 28 days beyond discontinuation of study treatment.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | From screening until disease progression or discontinuation of study
Time to progression (TTP) | From screening until disease progression or discontinuation of study
Duration of response (DR) | From screening until disease progression or discontinuation of study
Overall survival (OS) | From screening until disease progression or discontinuation of study
Probability of survival at 1 year | From screening until disease progression or discontinuation of study

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (13):
- United States (10):
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, City of Saint Peters, Missouri
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, Chapel Hill, North Carolina
  - Pfizer Investigational Site, Clinton, North Carolina
  - Pfizer Investigational Site, Goldsboro, North Carolina
  - Pfizer Investigational Site, Pollocksville, North Carolina
  - Pfizer Investigational Site, Wilson, North Carolina
  - Pfizer Investigational Site, Pittsburgh, Pennsylvania
  - Pfizer Investigational Site, Charlottesville, Virginia
- Pfizer Investigational Site, Orbassano (Torino), Italy
- Spain (2):
  - Pfizer Investigational Site, Badalona, Barcelona
  - Pfizer Investigational Site, Barcelona, BARCELONA

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6181040&StudyName=Study%20Of%20SU011248%20In%20Patients%20With%20Metastatic%20Non-Small%20Cell%20Lung%20Cancer%20%20